CLINICAL TRIAL: NCT04648683
Title: Postoperative Telehealth Mindfulness Intervention to Improve Pain-related Outcomes and Reduce Opioid Use After Lumbar Spine Surgery
Brief Title: Postoperative Telehealth Mindfulness Intervention After Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Carrie Brintz, Assistant Professor, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201486; K23AT011569 (NIH)
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Results first posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Chronic Low-back Pain; Postsurgical Pain; Opioid Use; Lumbar Spine Surgery
Keywords: Mindfulness; Telehealth; Mindfulness-based intervention
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Two-arm, nonrandomized, repeated measures design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual telehealth mindfulness (Experimental): Telehealth mindfulness sessions delivered one-on-one with mindfulness therapist
  Interventions: Behavioral: Individual telehealth mindfulness
- Group Telehealth Mindfulness (Experimental): Telehealth mindfulness sessions delivered in a small-group format with mindfulness therapist
  Interventions: Behavioral: Group telehealth mindfulness

INTERVENTIONS:
Behavioral: Individual telehealth mindfulness — Participants who enroll and complete lumbar spine surgery will participate in a one-on-one telehealth-delivered (online with audio and video) mindfulness intervention with a trained mindfulness therapist. The intervention is adapted from mindfulness-based cognitive therapy and includes eight, weekly sessions lasting 75 minutes each (except the first session which lasts 90 minutes).
  Arms: Individual telehealth mindfulness
Behavioral: Group telehealth mindfulness — Participants who enroll and complete lumbar spine surgery will participate in a group-delivered telehealth (online with audio and video) mindfulness intervention with a trained mindfulness therapist. The intervention is adapted from mindfulness-based cognitive therapy and includes eight, weekly sessions lasting 90 minutes each.
  Arms: Group Telehealth Mindfulness

SUMMARY:
Lumbar spine pain is the leading cause of years lived with a disability and affects over 50 million individuals in the United States. Rates of spine surgeries performed to address degenerative spine conditions have increased markedly. A subset of patients experience poor pain, functional, or quality of life outcomes after surgery.

This study will adapt and evaluate the feasibility and potential benefits of both a one-on-one and a group-delivered, face-to-face telehealth, mindfulness intervention for patients recovering from lumbar spine surgery. The goals of the intervention are to improve short and long-term pain management, reduce the need for long-term pain medications, and improve physical and psychological well-being after surgery. The study will result in a refined intervention manual based on feasibility, participant exit interviews and satisfaction surveys which will be piloted in a future randomized controlled trial.

DETAILED DESCRIPTION:
We will conduct a two-arm, nonrandomized, mixed-methods trial to refine a telehealth mindfulness-based intervention (MBI) for patients recovering from spine surgery. The procedures will be as follows:

1. Recruit, consent and enroll up to 26 patients over a period of 8 months who are planning to have their first lumbar spine surgery for a degenerative spine condition at the Vanderbilt Comprehensive Spine Center. Recruitment will occur at a routine preoperative clinic visit or over the phone, with the spine surgeon's permission to approach the patient.
2. Two weeks after enrolled patients complete surgery, they will meet with an interventionist for eight, weekly one-on-one or group-delivered telehealth MBI sessions over a Zoom online telehealth platform. Sessions will be 75 minutes long (90 minutes for the first session). Sessions will be audio recorded and the interventionists will be supervised weekly.
3. Participants will complete self-report assessments prior to surgery, two weeks after surgery (pre-intervention) and three months after surgery (post-intervention).
4. After completing the intervention, participants will complete an intervention satisfaction survey and an audio-recorded 30-minute semi-structured interview over the phone to provide feedback regarding their experience with the intervention components and relevance to their postoperative recovery.
5. We will code and analyze interview data continuously (every 2-4 interviews) until we reach data saturation and then integrate results from interviews and self-report surveys to determine relevant intervention adaptations, constructing a refined intervention protocol for pilot testing in a randomized controlled trial. We anticipate needing approximately 13-20 participants to complete interviews to reach data saturation (i.e. no new, relevant information obtained from interviews).

ELIGIBILITY:
Inclusion criteria:

1. English-speaking adults
2. Between the ages of 18 and 90
3. Scheduled for a laminectomy and/or fusion at Vanderbilt Spine Center
4. Scheduled for their first lumbar spine surgery
5. Radiographic evidence of a degenerative condition including but not limited to spinal stenosis, spondylosis with or without myelopathy, and spondylolisthesis
6. Presence of back and/or lower extremity pain persisting for at least 3 months
7. Access to stable internet.
8. Able to participate in weekly, remote sessions with a study therapist for 8 weeks after surgery

Exclusion criteria:

1. Microsurgical technique as the primary procedure (i.e. isolated laminotomy or microdiscectomy)
2. Having surgery for the primary indication of a spinal deformity
3. Having surgery secondary to pseudarthrosis, trauma, infection, or tumor
4. Current/history of a primary psychotic or major thought disorder or hospitalization for reasons related to psychosis
5. Diagnosis of Alzheimer's disease or another form of dementia
6. Traumatic Brain Injury (greater than mild severity)
7. History of bipolar disorder or dissociative disorder
8. Active substance use disorder (in past month)
9. Current Posttraumatic Stress Disorder (PTSD) symptoms (in past month)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie E Brintz, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Spine Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Individual Telehealth Mindfulness | Group Telehealth Mindfulness
Started | 10 | 0
Completed | 3 | 0
Not Completed | 7 | 0

BASELINE CHARACTERISTICS:
Population: The group arm of the study was discontinued due to difficulty enrolling enough participants for a group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Individual Telehealth Mindfulness | Group Telehealth Mindfulness | Total
Number analyzed (Participants) | 10 | 0 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (16.6) |  | 62.3 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  | 3
  Male | 7 |  | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 10 |  | 10
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 2 |  | 2
  White | 5 |  | 5
  More than one race | 0 |  | 0
  Unknown or Not Reported | 2 |  | 2
Education [Count of Participants; unit: Participants]
  High School diploma or GED | 3 |  | 3
  Two- or Four-year college degree | 3 |  | 3
  Post-college | 2 |  | 2
  Unknown or not reported | 2 |  | 2
Employment [Count of Participants; unit: Participants]
  Employed and currently working | 2 |  | 2
  Employed but not working (short-term disability or leave) | 2 |  | 2
  Unemployed | 3 |  | 3
  Unknown or not reported | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - Study Retention
Description: Percentage of participants enrolled who complete the study
Time Frame: 3 months following lumbar spine surgery
Population: Group arm discontinued
Measure: Count of Participants; unit: Participants
Arm/Group | Individual Telehealth Mindfulness | Group Telehealth Mindfulness
Number analyzed (Participants) | 10 | 0
Participants | 3 |

2. Primary Outcome: Feasibility - Session Attendance
Description: Percent of sessions attended out of 8
Time Frame: 3 months following lumbar spine surgery
Population: 5 participants started intervention. Remaining 5 participants withdrew prior to starting intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Individual Telehealth Mindfulness | Group Telehealth Mindfulness
Number analyzed (Participants) | 5 | 0
Participants
  8 sessions | 3 |
  3 sessions | 1 |
  1 session | 1 |

3. Primary Outcome: Acceptability - Satisfaction With Intervention
Description: Nine items assessing satisfaction with the postsurgical telehealth mindfulness intervention (sum of item scores; higher scores indicate higher satisfaction; scores can range from 7 to 55)
Time Frame: 3 months following lumbar spine surgery
Population: Group arm discontinued
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individual Telehealth Mindfulness | Group Telehealth Mindfulness
Number analyzed (Participants) | 3 | 0
score on a scale | 53.0 (2.0) |

4. Secondary Outcome: Pain Bothersomeness
Description: One item assessing how bothersome pain has been in the past 7 days from not at all = 0 to extremely = 4. A higher scores indicates higher pain bothersomeness.
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Individual Telehealth Mindfulness
Number analyzed (Participants) | 3
units on a scale | 0.3 (0.6)

5. Secondary Outcome: Pain Interference Short-form 4a
Description: Pain Interference short-form 4a from the Patient Reported Outcomes Measurement Information System scale. Measures interference of pain in day to day activities, work around the home, participation in social activities, and household chores over the past 7 days. Raw scores are converted to T-scores with a population mean of 50 and standard deviation of 10. A lower T-score indicates lower pain interference, or a better outcome.
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Individual Telehealth Mindfulness
Number analyzed (Participants) | 3
T-score | 46.3 (8.1)

6. Secondary Outcome: Overall Pain Intensity
Description: 1 item from the Patient Reported Outcomes Measurement Information System (PROMIS), with average pain intensity over the past 7 days rated on 0-10 scale with lower values indicating less pain, or better outcome.
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Individual Telehealth Mindfulness
Number analyzed (Participants) | 3
units on a scale | 0.7 (0.6)

7. Secondary Outcome: Back and Leg Pain Intensity
Description: 2 items assessing back and leg pain intensity on a scale of 0-10 over the past 7 days, described as pain when off medication or medication has worn off. Lower scores indicate less pain, or better outcome.
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Individual Telehealth Mindfulness
Number analyzed (Participants) | 3
units on a scale
  Back pain | 0.7 (0.6)
  Leg Pain | 0.3 (0.6)

8. Secondary Outcome: Self-reported Opioid Medication Use
Description: Measured as average number of opioid pills per day (name and dose specified) and converted to morphine equivalent dose.
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: milligrams of morphine equivalents
Arm/Group | Individual Telehealth Mindfulness
Number analyzed (Participants) | 3
milligrams of morphine equivalents | 0.0 (0.0)

9. Secondary Outcome: Anxiety Short Form 4a
Description: Anxiety short-form 4a - Patient Reported Outcomes Measurement Information System. 4 items assessing anxiety symptoms in the past 7 days (e.g. "I felt fearful"). Raw scores are converted to T-scores with a population mean of 50 and standard deviation of 10. Lower scores represent lower anxiety, a better outcome.
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Individual Telehealth Mindfulness
Number analyzed (Participants) | 3
T-score | 40.3 (0.0)

10. Secondary Outcome: Depression Short Form 4a
Description: Depression short-form 4a - Patient Reported Outcomes Measurement Information System scale. 4 items assessing depressive symptoms over the past 7 days (e.g. "I felt worthless). Raw scores are converted to T-scores with a population mean of 50 and standard deviation of 10. A lower score indicates less depression, a better outcome.
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Individual Telehealth Mindfulness
Number analyzed (Participants) | 3
T-score | 43.6 (4.6)

11. Secondary Outcome: Oswestry Disability Index
Description: Assesses impact of pain on level of functioning in 10 areas (e.g. walking, sleep, social life). Scores range from 0-100. Lower scores indicate lower level of disability due to pain, a better outcome.
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individual Telehealth Mindfulness
Number analyzed (Participants) | 3
score on a scale | 18.0 (19.1)

12. Secondary Outcome: Pain Catastrophizing Scale
Description: 13 items assessing thoughts and feelings when in pain (e.g. "I become afraid that the pain will get worse." Scores range from 0-52. Lower scores indicate lower pain catastrophizing, a better outcome.
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individual Telehealth Mindfulness
Number analyzed (Participants) | 3
score on a scale | 1.3 (2.3)

13. Secondary Outcome: Pain Self-efficacy Questionnaire
Description: 10 items assessing confidence in ability to do certain things despite pain (e.g. "I can enjoy things, despite the pain." Scores range from 0 to 60. Higher scores indicate greater pain self-efficacy, a better outcome.
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individual Telehealth Mindfulness
Number analyzed (Participants) | 3
score on a scale | 52.7 (12.7)

14. Secondary Outcome: Perceived Stress Scale - 4
Description: 4 items assessing perceived level of stress in the past month (e.g. "In the last month, how often have you felt that you were unable to control the important things in your life?"). Scores range from 0-16. Lower scores indicate lower perceived stress, a better outcome.
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individual Telehealth Mindfulness
Number analyzed (Participants) | 3
score on a scale | 4.0 (4.0)

15. Secondary Outcome: Tampa Scale for Kinesiophobia -13
Description: 13 items assessing fear of movement (e.g. "I'm afraid that I might injure myself if I exercise." Scores range from 13-52. Lower scores indicate lower levels of kinesiophobia, a better outcome.
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individual Telehealth Mindfulness
Number analyzed (Participants) | 3
score on a scale | 24.5 (8.4)

16. Secondary Outcome: Five Facet Mindfulness Questionnaire - 15
Description: 15 items assessing 5 facets of mindfulness, including observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Scores range from 1 to 5 (calculated by taking the average of the total sum score). Higher scores indicate higher levels of mindfulness, a better outcome.
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individual Telehealth Mindfulness
Number analyzed (Participants) | 3
score on a scale | 3.8 (0.5)

ADVERSE EVENTS:
Time Frame: From enrollment (prior to surgery) to 3 months after spine surgery, up to 4 months.
Description: Adverse events collected if they were reported by participants.
Arm/Group | Individual Telehealth Mindfulness
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT04648683/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT04648683/ICF_002.pdf